CLINICAL TRIAL: NCT00810810
Title: Immunomodulation Following Transfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Bloodworks (Other)
Responsible Party: Principal Investigator, Karen Nelson, Director, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29792; 1P50HL081015 (NIH)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Blood Component Transfusion
Keywords: Blood Component Transfusion; Leukoreduction; HLA antibody; Immunosuppression
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Intervention Model Description: Individuals who consented for study were scheduled for cardiac surgery. They were randomized to one of three arms to receive blood components prepared by different, but clinically acceptable processes. If they required transfusion from 2 days prior to surgery until 30 days post surgery they received study product. Blood samples were collected prior to surgery and at two points after surgery.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical teams caring for patients were not masked. Laboratory personnel were masked until all testing completed.
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Blood components with no additional treatment
  Interventions: Biological: Standard blood components
- 2 (Experimental): Blood components leukoreduced
  Interventions: Biological: Leukoreduced blood components
- 3 (Experimental): Blood components leukoreduced and irradiated
  Interventions: Biological: Leukoreduced and irradiated

INTERVENTIONS:
Biological: Standard blood components — Transfusion, if ordered by physician, with unfiltered red blood cells and apheresis platelets
  Arms: 1
Biological: Leukoreduced blood components — Transfusion, if ordered by a physician, of leukoreduced red blood cells and apheresis platelets
  Arms: 2
Biological: Leukoreduced and irradiated — Transfusion, if ordered by physician, of gamma irradiated leukoreduced red blood cells and gamma irradiated apheresis platelets
  Arms: 3

SUMMARY:
This study is designed to provide information on patients' immune response after exposure to transfused blood.

Blood transfusions may have opposite immune effects on patients. One is sensitization. The other is immunosuppression. The magnitude of these effects in patients who are not on chemotherapy is unknown.

These effects are thought to be due largely to white blood cells present in the transfusion product. "Leukofiltration" and "gamma-irradiation" are the special treatments that deplete white blood cells. A combination of leukofiltration and gamma-irradiation pretreatment of donor blood is thought to deplete the white blood cells most effectively.

In this study, patients scheduled for cardiac surgery are randomly assigned to receive blood products pretreated in one of three ways: untreated, filtered or filtered and irradiated. If their physician orders transfusions, they will receive products assigned to their group. Patients are asked to provide two blood samples during the 4 weeks after surgery.

Studies will measure changes in antibody to HLA and in cells that regulate the immune response. The levels of sensitization and immunosuppression will be correlated to the transfusion products received.

DETAILED DESCRIPTION:
Blood transfusions may have opposite immune effects on patients. One is sensitization. The other is immunosuppression. The magnitude of this problem in patients who are not on chemotherapy is unknown.

Of patients who do receive donor blood, 50-90 percent become sensitized (make antibody) to HLA proteins present on white blood cells in the donor blood. This is an undesired effect in patients who need an organ or stem cell transplant, as it increases the risk of rejection. Another effect of receiving a blood transfusion, immunosuppression, causes a decreased immune response that compromises patients' ability to fight off infection or tumor cells.

These effects - sensitization and immunosuppression - are thought to be due largely to white blood cells present in the transfusion product. Doctors order specially pretreated blood transfusions that have been depleted of white blood cells with the aim of minimizing risks in an "immunocompromised" patient. "Leukofiltration" and "gamma-irradiation" are the special treatments that deplete white blood cells. A combination of leukofiltration and gamma-irradiation pretreatment of donor blood is thought to deplete the white blood cells most effectively. Therefore, blood is pretreated both ways before it is given to patients who need a stem cell transplant or others who are immunosuppressed.

Sometimes the pretreated leukofiltration and gamma-irradiated blood is used for "regular" patients who are not immunocompromised so the blood is used before it expires and not wasted. However, doctors do not know for sure whether these expensive pretreatments are really beneficial for "regular" patients such as those undergoing cardiac surgery and whether they would change the risk of developing sensitization or immunosuppression.

In this study, patients are randomly assigned to receive blood products pretreated in one of three ways: untreated, filtered or filtered and irradiated. If their physician orders transfusions, they will receive products assigned to their group. Patients are asked to provide two blood samples during the 4 weeks after surgery. Studies will measure changes in antibody to HLA and in cells that regulate the immune response.

It is unknown which treatment (leukofiltration with or without gamma-irradiation compared to no pretreatment) is most beneficial in patients who are not immunosuppressed.

This study is designed to provide information on patients' immune response after exposure to transfused blood. This information may be useful to caring for patients in the future who require transfusion for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 year of age
* Scheduled for open heart surgery of cardiopulmonary bypass that involves: CABG, CABG with valve, aneurysm repair
* Urgent or elective surgery

Exclusion Criteria:

* Scheduled for open heart surgery of cardiopulmonary bypass that involves: placement of a ventricular assist device, cardiac transplantation, aortic dissection repair
* Emergent surgery
* participation in other clinical research studies within 30 days of randomization.
* Immunosuppressive treatment.
* Refuse blood transfusion
* Disease or condition placing subject at undue risk or decision of attending doctor.
* Condition requiring high volume transfusion therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Nelson, PhD, Principal Investigator — Bloodworks; Gabriel Aldea, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Nelson KA, Aldea GS, Warner P, Latchman Y, Gunasekera D, Tamir A, Gernsheimer T, Bolgiano D, Slichter SJ. Transfusion-related immunomodulation: gamma irradiation alters the effects of leukoreduction on alloimmunization. Transfusion. 2019 Nov;59(11):3396-3404. doi: 10.1111/trf.15555. Epub 2019 Oct 13. PMID 31608454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for cardiac surgery at the U. Washington or an affiliated program at Northwest Hospital had the study explained to them by the clinical team including a clinical research coordinator and consent was obtained.
  Recruitment began in August of 2006 and extended until August of 2010.
Pre-assignment Details: There were 7 individuals who consented but were not randomized: late discovery of exclusionary criteria, surgery cancelled, individual withdrew.
Groups:
- 4. No Transfusion: This arm includes participants from arms 1, 2 and 3 who did not require nor receive transfusions of red blood cells or platelets while they were on study. These participants were moved to this arm after study completion, prior to analysis.
- 1. Standard: Patients received unfiltered red blood cells and apheresis platelets if transfusions were ordered by their providers while on study (2 days prior to surgery to 30 days post surgery).
- 2. Leukoreduced: Patients received filter leukoreduced red blood cells and apheresis platelets collected leukoreduced if transfusions were ordered by their providers while on study (2 days prior to surgery to 30 days post surgery).
- 3. Leukoreduced Gamma Irradiated: Patients received filter leukoreduced red blood cells that were gamma irradiated and apheresis platelets collected leukoreduced and gamma irradiated if transfusions were ordered by their providers while on study (2 days prior to surgery to 30 days post surgery).
Period: Overall Study
Arm/Group | 4. No Transfusion | 1. Standard | 2. Leukoreduced | 3. Leukoreduced Gamma Irradiated
Started | 124 | 49 | 56 | 51
Completed | 124 | 38 | 45 | 38
Not Completed | 0 | 11 | 11 | 13
Not completed — Withdrawal by Subject | 0 | 8 | 10 | 8
Not completed — Physician Decision | 0 | 3 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4. No Transfusion | 1. Standard | 2. Leukoreduced | 3. Leukoreduced Gamma Irradiated | Total
Number analyzed (Participants) | 124 | 38 | 45 | 38 | 245
Age, Customized [Count of Participants; unit: Participants]
  18 Years and older | 124 | 38 | 45 | 38 | 245
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data on sex/gender was not recorded as neither the primary nor the secondary outcomes used those measures in the analysis.
  All patients presenting to the service who did not have one or more exclusionary criteria were approached for consent to the study.
  Participants
    unknown | 124 | 38 | 45 | 38 | 245
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 124 | 38 | 45 | 38 | 245

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in the Production of Antibody to HLA Antigens
Description: Blood samples were collected prior to surgery and at two times after surgery. Serum was tested for the presence of IgG antibody to HLA. the results of the samples collected after surgery were compared to those in the sample collected prior to surgery.
Time Frame: 0 to 5 weeks after surgery
Population: Antibody tests were invalid for some participants in Arm 1. Their sera contained interfering substances.
Measure: Count of Participants; unit: Participants
Arm/Group | 4. No Transfusion | 1. Standard | 2. Leukoreduced | 3. Leukoreduced Gamma Irradiated
Number analyzed (Participants) | 124 | 38 | 45 | 38
Participants
  Baseline antibody negative, antibody increased: number analyzed (Participants) | 79 | 20 | 25 | 23
  Baseline antibody negative, antibody increased | 2 | 6 | 2 | 5
  Baseline antibody positive, antibody increased: number analyzed (Participants) | 44 | 13 | 20 | 15
  Baseline antibody positive, antibody increased | 11 | 10 | 10 | 8

2. Secondary Outcome: Number of Participants With Changes in the Number or Cytokine Profile of CD4 T Regulatory Cells or NKT Cells. Number of Participants With Changes in Numbers of Cells Producing TGFB1. Number of Participants With Changes in Secretion of Cytokines
Description: Blood samples were collected prior to surgery and at two times after surgery. White blood cells were isolated and frozen. The thawed cells were tested for the numbers and phenotype of regulatory cells and for the production of regulatory cytokines. Results obtained from samples collected after surgery were compared to the results obtained from the sample collected prior to surgery.
Time Frame: 0 to 5 weeks after surgery
Population: The study used stringent criteria for acceptance of these cellular assays. Invalid tests were not included in the analysis, therefor the numbers reported in the Outcome Measures table do not add up to the number analyzed for each test.
Measure: Count of Participants; unit: Participants
Arm/Group | 4. No Transfusion | 1. Standard | 2. Leukoreduced | 3. Leukoreduced Gamma Irradiated
Number analyzed (Participants) | 71 | 20 | 25 | 23
Participants
  Number of MNC producing TGFB1: number analyzed (Participants) | 67 | 18 | 23 | 19
  Number of MNC producing TGFB1: Increased | 30 | 11 | 12 | 7
  Number of MNC producing TGFB1: Not increased | 37 | 7 | 11 | 12
  Number of CD4+ IL4+ iNKT cells: number analyzed (Participants) | 70 | 19 | 25 | 23
  Number of CD4+ IL4+ iNKT cells: Increased | 22 | 10 | 15 | 4
  Number of CD4+ IL4+ iNKT cells: Not increased | 48 | 9 | 10 | 19
  Number of CD4+ IFNg+ iNKT cells: number analyzed (Participants) | 70 | 19 | 25 | 23
  Number of CD4+ IFNg+ iNKT cells: Increased | 9 | 1 | 2 | 1
  Number of CD4+ IFNg+ iNKT cells: Not increased | 61 | 18 | 23 | 22
  Number of CD4- IL4+ iNKT cells: number analyzed (Participants) | 70 | 19 | 25 | 23
  Number of CD4- IL4+ iNKT cells: Increased | 17 | 1 | 2 | 1
  Number of CD4- IL4+ iNKT cells: Not increased | 53 | 18 | 23 | 22
  Number of CD4- INFg+ iNKT cells: number analyzed (Participants) | 70 | 19 | 25 | 23
  Number of CD4- INFg+ iNKT cells: Increased | 13 | 1 | 1 | 2
  Number of CD4- INFg+ iNKT cells: Not increased | 57 | 18 | 24 | 21
  IL-10 produced by PBMC: number analyzed (Participants) | 71 | 19 | 23 | 23
  IL-10 produced by PBMC: Increased | 45 | 14 | 16 | 8
  IL-10 produced by PBMC: Not increased | 26 | 5 | 7 | 15
  CD4+Number of CD25+FoxP3+ T cells: number analyzed (Participants) | 64 | 20 | 24 | 20
  CD4+Number of CD25+FoxP3+ T cells: Increased | 5 | 7 | 9 | 4
  CD4+Number of CD25+FoxP3+ T cells: Not increased | 59 | 13 | 15 | 16
  Number of CD4+CD25+CTLA4+ T cells: number analyzed (Participants) | 64 | 20 | 24 | 20
  Number of CD4+CD25+CTLA4+ T cells: Increased | 8 | 9 | 11 | 3
  Number of CD4+CD25+CTLA4+ T cells: Not increased | 56 | 11 | 13 | 17

ADVERSE EVENTS:
Time Frame: Duration on study - 30 days post surgery.
Description: The only study related adverse event would have been due to the phlebotomy to collect study blood samples and none were reported.
  Participants received transfusion therapy as ordered by their clinical team. None of the blood products were experimental.
Arm/Group | 4. No Transfusion | 1. Standard | 2. Leukoreduced | 3. Leukoreduced Gamma Irradiated
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/49 | 0/56 | 0/51
Other Adverse Events (participants affected / at risk) | 0/124 | 0/49 | 0/56 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No